CLINICAL TRIAL: NCT06841289
Title: The Effect of Pediatric Invasive Pictorial Shield (PIPS) and Distraction Card Use on Pain, Fear and Anxiety in Blood Collection Procedure
Brief Title: The Effect of Pediatric Invasive Pictorial Shield (PIPS) and Distraction Card Use in Blood Collection Procedure
Acronym: PIPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dilek Kucuk Alemdar (Other)
Responsible Party: Sponsor-Investigator, Dilek Kucuk Alemdar, Professor, Ordu University
Organization: Ordu University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: KAEK360
Record Dates: First submitted 2025-02-18; First posted 2025-02-24 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Pain Management; Fear Anxiety; Child
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Intervention Model Description: The study was a randomized controlled experimental, prospective study.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: After the children who met the inclusion criteria were assigned to the study groups by stratified block randomization, their written informed consent will be obtained through the informed consent form without informing their parents which group they are included in. Since the researcher will administer the PIPS and distraction cards to the children, blinding will not be possible. However, in order to prevent detection bias, the output measurements of the study will be made by the nurse working in the blood collection unit where the study will be conducted, who does not know who is in the experimental group and who is in the control group. In order to prevent bias in the evaluation of the data, the study groups will be coded in the database as A, B and C by someone other than the researcher, and the data be analyzed by a statistical expert independent of the research. It was aimed to prevent statistical and reporting bias by blinding in terms of output measurements, statistical analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pediatric Invasive Pictorial Shield (PIPS) (Experimental): It is a device used to distract children during clinical procedures (blood sampling, invasive procedures, etc.) by making them feel less pain, stress and fear. It is an 18x15 cm 3D printed device designed to be worn around the upper arm, above the elbow, and used to hide the procedure from view and attract the child's attention with stickers printed on one side.
  Interventions: Combination Product: Pediatric Invasive Pictorial Shield (PIPS)
- Distraction cards (Other): Distraction cards consist of picture cards with various hidden pictures and patterns. These hidden pictures and patterns can only seen by the child if he/she looks carefully. During the procedure, the child is expected to focus on the cards and answerabout the pictures and shapes on the cards. In this study, 5X8 cm cards with various pictures and shapes will be used . For the children in this group, the pain, fear will be scored 1 minute before, during and 1 minute after the blood collection procedure.
  Interventions: Behavioral: Distraction cards
- Control (No Intervention): No distraction method will be applied to the children in the control group before the blood collection procedure. After explaining the procedure according to the developmental level of the child, blood collection will be performed by the same nurse in accordance with the institutional policy.

INTERVENTIONS:
Combination Product: Pediatric Invasive Pictorial Shield (PIPS) — It is a device used to distract children during clinical procedures (blood sampling, invasive procedures, etc.) by making them feel less pain, stress and fear. It is an 18x15 cm 3D printed device designed to be worn around the upper arm, above the elbow, and used to hide the procedure from view and attract the child's attention with stickers printed on one side. The device is fixed on the child's arm by means of a tourniquet that can be interchangeably attached. The child asked questions about the pictures related to the stickers to distract his/her attention from the procedure. While answering these questions, the child will not see the procedures and will pay attention to the pictures, while the procedural procedure (such as blood sampling, intravenous intervention) will be performed. For the children in this group, the pain, fear will be scored 1 minute before, during and 1 minute after the blood collection procedure.
  Arms: Pediatric Invasive Pictorial Shield (PIPS)
Behavioral: Distraction cards — Distraction cards consist of picture cards with various hidden pictures and patterns. These hidden pictures and patterns can only seen by the child if he/she looks carefully. During the procedure, the child is expected to focus on the cards and answerabout the pictures and shapes on the cards. In this study, 5X8 cm cards with various pictures and shapes will be used.
  Arms: Distraction cards

SUMMARY:
This study was planned as a randomized controlled experimental study to minimize the pain, anxiety and fear of the child during venous blood sampling in order to avoid a painful experience in the future. The research will be conducted in the Pediatric Blood Collection Unit of Giresun Gynecology and Obstetrics Training and Research Hospital in children aged 6-10 years. The research data will be collected using the "Information Form on Descriptive Characteristics of the Child and Blood Collection Procedure, Child Anxiety Scale-Disposition (CAS-D), Oucher Scale, Child Fear Scale (CFS), Venham Pictorial Anxiety Scale (VRAAS)" and Nurse-Patient Cooperation and Parent Satisfaction Form (NPPS-EMF).

DETAILED DESCRIPTION:
Invasive procedures are the most common and important sources of pain, anxiety, stress and fear for children. Painful procedures also cause reluctance to medical procedures and distrust of nurses in both children and parents. Pain, anxiety and fear from needle procedures in childhood can persist into adulthood. It may cause negative emotional effects in the long term. Therefore, it is very important to reduce or eliminate pain during stressful and uncomfortable procedures in children. Nurses should also provide atraumatic care to children by minimizing pain. Eliminating pain and improving the quality of life of children should be one of the main goals of nursing care. The methods used in pain control in children are pharmacologic and nonpharmacologic methods. One of the non-pharmacologic methods, the technique of distraction, is the concentration of attention on a stimulus other than pain. Unlike what we have previously encountered in the literature, the Pediatric Invasive Pictorial Shield (PIPS) also aims to minimize the impact of the intervention by preventing the child from seeing the procedure being performed. Distraction cards are also known to be an effective method in children. This study was planned as a randomized controlled experimental study to minimize the pain, anxiety and fear of the child during venous blood sampling in order to avoid a painful experience in the future. The research will be conducted in the Pediatric Blood Collection Unit of Giresun Gynecology and Obstetrics Training and Research Hospital in children aged 6-10 years. The research data will be collected using the "Information Form on Descriptive Characteristics of the Child and Blood Collection Procedure, Child Anxiety Scale-Disposition (CAS-D), Oucher Scale, Child Fear Scale (CFS), Venham Pictorial Anxiety Scale (VRAAS)" and Nurse-Patient Cooperation and Parent Satisfaction Form (NPPS-EMF).

ELIGIBILITY:
Inclusion Criteria:

* The child must be between 6-10 years old, and the child and parents must agree to participate in the study
* Blood collection is done by the same nurse
* Standard information is given to the child and family before blood collection - - The blood collection method to be used for the procedure (butterfly set
* Children should have the perception level to evaluate the pain/fear/anxiety scale (successfully complete the scale tests)
* The child does not have any auditory, mental or neurological disability that may affect the child's participation in the research
* The child has no hearing, speech or visual impairment Blood collection from the antecubital region
* Single attempt intervention.

Exclusion Criteria:

* The child has any special needs (physical, sensory or mental)
* The child is admitted to the hospital with a complaint of acute pain
* Body temperature outside the range of 36.5-37.2°C153
* Having a disease that can cause chronic pain The child has taken analgesics in the last 6 hours
* The child has a health problem that may affect the level of pain (tissue trauma, burn, fracture, etc.).

Ages: 6 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2025-02-17 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-06-15 (Actual)

PRIMARY OUTCOMES:
Oucher Scale | 1 minute before, during procedure and 1 minute after the blood collection procedure.
  Oucher is a poster-like tool designed to help children self-report the intensity of their pain. The Oucher consists of two scales: a numerical scale from 0-10 for older children and a photographic scale with six pictures for younger children. The Oucher can be used to assess pain intensity whenever the child is awake and conscious. Oucher can be used in children aged 3-12 years.
Child Anxiety Scale-Dispositional (CAS-D) | 1 minute before, during procedure and 1 minute after the blood collection procedure.
  The CAS-D is shaped like a thermometer with a bulb at the bottom and horizontal lines at intervals going upwards. In this scale for children aged four to ten, children instructed to "Imagine that all your anxious or nervous feelings are at the bulb or bottom of the thermometer". "If you are a little worried or nervous, the emotions might go up a little on the thermometer. If you are very, very anxious or nervous, emotions all the way to the top. Put a line on the thermometer showing how anxious or nervous you are". To measure state anxiety (CAS-D), the child is asked to mark how they feel "right now". The score can vary between 0 and 10
Child Fear Scale (CFS) | 1 minute before, during procedure and 1 minute after the blood collection procedure.
  This scale is used to determine the child's level of fear. The child fear scale is a visual scale consisting of five facial expressions characterized as no reaction (0=no anxiety) and scared face (4=severe anxiety) and can be scored from 0 to 4. It is intended for children aged 5-10 years (Gerçeker et al., 2018)
Venham Pictorial Anxiety Scale (VRAQ) | 1 minute before, during procedure and 1 minute after the blood collection procedure.
  It was developed as a situational anxiety scale for children. It measures anxiety appropriate for children in stressful situations. The scale was developed by Venham et al. in 1979. The scale is used for children over 3 years of age. The scale consists of eight sections and each section two pictures. The pictures in each section are shown to the child in order. The picture with anxiety is given 1 point and the picture without anxiety is 0 point. The lowest score is 0 and the highest score is 8 points. In the scoring system from 0 to 8, as the number of points increases, the rate of anxiety increases

SECONDARY OUTCOMES:
Nurse-Patient Collaboration and Parental Satisfaction Form (NPPC-EMF) | 5 minute after the blood collection procedure.
  Nurse-Patient Cooperation Level and Parental Satisfaction Form was developed by Aydemir in 2020. "Nurse-Patient Cooperationsection consists of two questions directed to the nurse who performed the procedure. The scope of the questioning includes rating how the patient's compliance is during the application process and whether the continuity of the application is desired. The patient is asked to rate the patient's compliance with the procedure between zero and 10 points. Zero is the worst and 10 the best compliance. The status of wanting the application again was graded with the responses of I would like, I am undecided and I do not want. In the "Satisfaction of the Patient's Parent" section, there are two questions directed to the parents regarding the satisfaction and continuity of the application. Parental satisfaction was scaled on a five-point Likert scale one to five, with one being the most dissatisfied

CONTACTS AND LOCATIONS:
Overall Officials: Dilek Küçük Alemdar, Professor, Study Director — Ordu University
Locations (1):
- Ordu Üniversitesi, Ordu, Ordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No